CLINICAL TRIAL: NCT00739856
Title: Efficacy of ECT in Chronic, Severe, Antidepressant- And CBT-Refractory Posttraumatic Stress Disorder: An Open, Prospective Study
Brief Title: Use of Electroconvulsive Therapy (ECT) in Chronic, Severe, Treatment Resistant Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College Srinagar (Other Government)
Collaborators: Government Psychiatric Diseases Hospital, Srinagar (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMCPTSD_ECT2005
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; electroconvulsive therapy; medication refractoriness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Electroconvulsive Therapy — ECT was administered using the MECTA-SR1 apparatus. The current amplitude was 800 mA, pulse width was 1.5 ms, and pulse frequency was 50 Hz. Stimulus duration was increased as required to elicit an adequate seizure, defined as at least 25 s with EEG monitoring. The ECT course was fixed, and comprised 6 treatments administered with bitemporal electrode placement at a twice-weekly frequency

SUMMARY:
Post Traumatic Stress Disorder is a chronic debilitating illness and few treatment options have demonstrated effectiveness. The study will look at the use of electroconvulsive therapy for the treatment of Post Traumatic Stress disorder in patients who have not responded to multiple antidepressants or cognitive behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD
* Treatment resistance to 4 different antidepressants from 3 different classes
* Treatment resistance to CBT
* Severe PTSD

Exclusion Criteria:

* Significant substance abuse
* Pregnancy
* History of Traumatic Brain Injury
* Unstable comorbid medical illness
* Organic brain syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered Posttraumatic Stress Disorder Scale (CAPS) SCORE

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale score | baseline, 48 hrs post 3rd, 6th ECT

CONTACTS AND LOCATIONS:
Overall Officials: Mushtaq Margoob, MD, Principal Investigator — Government Medical College Srinagar
Locations (1):
- Government Hospital for Psychiatric Disease, Srinagar, Jammu and Kashmir, India

REFERENCES:
- [Derived] Margoob MA, Ali Z, Andrade C. Efficacy of ECT in chronic, severe, antidepressant- and CBT-refractory PTSD: an open, prospective study. Brain Stimul. 2010 Jan;3(1):28-35. doi: 10.1016/j.brs.2009.04.005. Epub 2009 May 27. PMID 20633428